CLINICAL TRIAL: NCT02322957
Title: A Phase 1 Study Investigating the Pharmacokinetics of FV-100 With and Without Ritonavir in Healthy Volunteers
Brief Title: A Study Investigating the Pharmacokinetics of FV-100 With and Without Ritonavir in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ContraVir Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: ContraVir (Unknown)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTRV-FV-1-008
Record Dates: First submitted 2014-12-15; First posted 2014-12-23 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Acute Herpes Zoster
MeSH Terms: interventions — FV-100

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Regimen A (Experimental): FV-100 400mg OD as a single dose fasted (>/= 8 hours)
  Interventions: Drug: FV-100
- Treatment Regimen B (Experimental): FV-100 400 mg OD as a single dose with ritonavir 200mg OD as a single fasted dose (>/= 8 hours)
  Interventions: Drug: FV-100

INTERVENTIONS:
Drug: FV-100 — Subjects will be randomized to one of two treatment sequences: AB or BA.

SUMMARY:
This study is designed to evaluate the potential for a PK drug-drug interaction between FV-100 and ritonavir. The study is a single-center, open-label, randomized, 2-way crossover design in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent
* Non-tobacco user for at least 3 months prior to selection
* Healthy on the basis of physical examination, medical history, ECG and clinical laboratory testing at screening

Exclusion Criteria:(must NOT meet the following)

* Infected with Hepatitis A, B, C, or HIV
* History of or any current medical condition which could impact safety of the participant
* A positive urine drug test
* Consumption of more than 2 units of alcoholic beverages per day or more than 14 per week
* Received an investigational drug or vaccine or used an investigational medical device within 3 months or 5 half-lives before the planned start of treatment or prior treatment with FV-100
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome(CYP) P450 enzymes and/or P-gp within 28 days prior to the first dose and throughout study
* Subjects who have, within 2 weeks prior to the first dose of study drug, ingested grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family or charbroiled meats

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The evaluation of safety of a single oral dose of FV-100 alone and when combined with a single oral dose of ritonavir | Two weeks
  Measuring the Cmax, Tmax and AUC for FV-100 pk profile
The evaluation of the pharmacokinetics of FV-100 and CF-1743 following a single oral dose of FV-100 administered alone and with a single oral dose of ritonavir | Two weeks
  Measuring the Cmax, Tmax and AUC for FV-100 pk profile when dosed with ritonavir